CLINICAL TRIAL: NCT06681909
Title: Adapting the Veggie Van Mobile Market Intervention to Address Disparities in Nutrition Security Among College Students
Brief Title: University At Buffalo Campus Veggie Van Mobile Market
Status: Active, not recruiting | Type: Observational
Sponsor: University at Buffalo (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Lucia A Leone, Principal Investigator, University at Buffalo
Other Study IDs: 1R21MD019367-01 (NIH); R21MD019367 (NIH)
Record Dates: First submitted 2024-11-06; First posted 2024-11-12 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-11

CONDITIONS: Food Habits; Food Selection
MeSH Terms: conditions — Feeding Behavior; Food Preferences

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Food Insecure Students: Undergraduate students who reported high to moderate food insecurity, are at least 18 years of age, speak English, and plan to return to the University at Buffalo campus in Spring 2025 will receive weekly fruit and vegetable incentives encouraging them to shop at the UB Veggie Van (intervention). They will complete incentivized data collection after 13 weeks of the intervention (incentives/access to UB Veggie Van).
  Interventions: Behavioral: UB Campus Veggie Van

INTERVENTIONS:
Behavioral: UB Campus Veggie Van — The UB Veggie Van is based on the Veggie Van, an evidence-based mobile produce market intervention. Mobile markets are like farmers' markets on wheels that travel to underserved communities selling high-quality, low-cost produce and healthy foods. The Veggie Van mobile market model was developed through multiple research studies on the efficacy, effectiveness, and implementation of the intervention, and is a multi-level intervention that addresses the five components of nutrition security (availability, accessibility, affordability, stability, and utilization). The UB Veggie Van is operated according to the Veggie Van model, with specific adaptations made to more effectively reach the campus community (Aim 1 of the larger funded study).
  Other Names: UB Veggie Van

SUMMARY:
The goal of this observational study is to develop an adaptable mobile produce market model to be used on college campuses to increase college students' access to fresh fruits and vegetables. Food insecurity on college campuses threatens academic success and student well-being, and affects first generation, lower-income, and racial/ethnic minority students at higher rates. This research will include a pilot campus mobile market operated on the University at Buffalo campus. The main questions it aims to answer are: 1.) What makes it hard for students to eat healthy foods on the University at Buffalo campus, 2.) How does a mobile market need to operate on a college campus to best reach students, and 3.) What is the relationship between mobile market use and changes in how many fruits and vegetables students eat, students' ability to consistently eat foods that promote health and well-being, and participation in the Special Nutrition Assistance Program (SNAP).

DETAILED DESCRIPTION:
As first-generation, low-income, and racial/ethnic minority students have improved their access to higher education, food insecurity in United States campuses has increased and threatens their academic success and well-being. College food pantries have been the most common solution but only offer short-term emergency relief, and stigma has prevented their use. To provide a longer-term evidence-based approach that honors students' choices and dignity, this research will inform the development of an adaptable campus mobile market model that consistently provides access to healthy food and promotes nutrition security. The clinical trial portion of the research will evaluate how intervention dosage, gauged by University at Buffalo Campus Veggie Van (UB Veggie Van) visits, total fruit and vegetable purchasing, and incentive redemption, is associated with changes in fruit and vegetable consumption (including skin carotenoids), nutrition security measures, and Special Nutrition Assistance Program (SNAP) enrollment from the beginning to the end of the semester.

ELIGIBILITY:
Inclusion Criteria:

* current students at the University at Buffalo
* completed the online campus survey (Aim 1 of larger funded project)
* experienced food insecurity during Spring 2024
* undergraduate students
* at least 18 years of age
* speak English
* must plan to return to the University at Buffalo campus in Spring 2025.

Exclusion Criteria:

* non-students
* non-English speaking
* students who will not return to campus in Spring 2025
* graduate students

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Food-insecure undergraduate students at the University at Buffalo in Buffalo, NY who are attending classes for the 2024-2025 school year.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2024-08-23 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Fruit and Vegetable Consumption | Collected at baseline and after the 13-week intervention period
  Fruit and vegetable consumption will be assessed using the 2021 Behavioral Risk Factor Surveillance System Fruit and Vegetable (FV) module
Nutrition Security | Collected at baseline and after the 13-week intervention period
  The Nutrition Security, Healthfulness Choice, and Dietary Choice Measure assesses factors associated with the ability of an individual to obtain foods that meet their nutritional and health needs and dietary preferences, without resource limitations or worry. Barriers to utilization will be assessed with a measure developed by Calloway et al., which includes eight items that assess tangible and intangible barriers to preparing healthful meals from the food a person can access.
Supplemental Nutrition Assistance Program (SNAP) Enrollment | Collected at baseline and after the 13-week intervention period
  A single survey question asking: "Did you participate in the following programs during the [semester before or during the intervention]?: Food stamps (Supplemental Nutrition Assistance Program or SNAP benefits), Special Supplemental Assistance Program for Women, Infants, and Children (WIC) benefits, Government cash assistance including Temporary Assistance for Needy Families (TANF), Social Security Insurance (SSI), Social Security Disability Insurance (SSDI), or government assistance (but not including social security benefits).

SECONDARY OUTCOMES:
Intervention Dosage | Collected throughout the 13-week intervention period
  Number of visits to the UB Veggie Van over the intervention period, total fruit and vegetable spending, and amount of purchasing incentives redeemed--these metrics will be tracked using the Veggie Van POS (Farmers Register).

OTHER OUTCOMES:
Process Measures | Collected after the 13-week intervention period
  Survey questions on the receipt and usage of the intervention and intervention materials, including newsletters, cooking demonstrations, recipes, educational materials, etc.
UB Campus Veggie Van Perceptions | Collected after the 13-week intervention period
  Measure student perceptions of the intervention using the Acceptability of Intervention Measure and the Intervention Appropriateness Measure.
Skin Carotenoids | Collected at baseline and after the 13-week intervention period
  We will use the "Veggie Meter", a noninvasive finger scan technology that relies on pressure-mediated reflection spectroscopy. Skin carotenoid measurements correlate positively and significantly with blood carotenoids and reported dietary intake.

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Leone, PhD, Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided